CLINICAL TRIAL: NCT04654247
Title: A Prospective, Single-center Study Evaluating the Effectiveness of Endo.Adm in Improving the Quality of Gastrointestinal Endoscopy
Brief Title: Endoscopic Quality Improvement System Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EA-19-004
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Adenoma Colon; Gastric Precancerous Condition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Endoscopists in control group were informed standard quality indicators requirements and the corresponding references during informed consent.
  Interventions: Behavioral: Control
- Feedback group (Experimental): Endoscopists in feedback group were informed standard quality indicators requirements and the corresponding references during informed consent. In addition to the quality requirements, endoscopists randomized to feedback group received customized quality reports feedback from Endo.Adm weekly.
  Interventions: Behavioral: Quality audit and feedback

INTERVENTIONS:
Behavioral: Quality audit and feedback — Endoscopists received quality report generated by Endo.Adm.
  Arms: Feedback group
Behavioral: Control — None feedback.
  Arms: Control group

SUMMARY:
We intend to develop intelligent quality control and management software based on the work of digestive endoscopic artificial intelligence in the Department of Gastroenterology, Wuhan University Renmin Hospital, to accurately and comprehensively assess the quality of gastrointestinal endoscopy and to provide a practical basis for improving the quality of digestive endoscopy in our endoscopic center.

ELIGIBILITY:
Inclusion Criteria:

Endoscopist:

1. Endoscopist with more than one year experience in gastrointestinal mirror operation;
2. Willing to further improve endoscopic quality through Endo.Adm feedback;
3. Ability to read, understand and sign informed consent; The investigator believes that the subject understands the flow of the clinical study and is willing and able to complete all research procedures and follow-up visits in conjunction with the research process.

Exclusion Criteria:

Endoscopist:

1. Have participated in other clinical trials;
2. Frequently attending in academic conference which is difficult to ensure the number of endoscopic operations;
3. Endoscopist who were either not present for both parts (phase1 and phase2) of the study.

Patients:

Colonoscopy:

1. Polyposis syndromes
2. Lumen obstruction
3. History of colorectal surgery
4. History of colorectal surgery

Gastroscopy:

1. Obstruction
2. History of gastric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 3 Months
  ADR was calculated by dividing the total number of patients being detected adenomas by the number of colonoscopies.
Gastric precancerous detection rate | 3 Months
  GPCs detection rate was calculated by dividing the total number of patients being detected gastric precancerous by the number of gastroscopies.

SECONDARY OUTCOMES:
Adcanced ADR | 3 months
  Adcanced ADR was calculated by dividing the total number of patients being detected ≥10mm in size, or adenomas with histopathology of tubulovillous, villous, adenocarcinoma, or high-grade dysplasia by the number of colonoscopies.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual de-identified participant data that underlie the results reported in this article and study protocol will be shared for investigators whose proposed use of the data has been approved by an independent review committee. Data can only be used to achieve aims in the approved proposal. Data disclosure begins 9 months and ends 36 months after article publication. To gain access, data requesters will need to sign a data access agreement. Proposals should be directed to the corresponding author.